

'Implementation and Validation of the Dutch Translation of the TAPS-tool: a Screener for Tobacco, Alcohol, Prescription Medication and Other Substances for Patients With Severe Mental Illness With and Without Intellectual Disabilities'

ECSW-2021-052

Date 07.04.2020



Region Regio Helmond - Peelland en Boekel

Department FACT

Adress Postbus 3, 5427 ZG BOEKEL

**Phone** 0492 - 84 43 00 **Date** 7 april 2020

Subject Participation on research on the TAPS-tool

## Dear sir / madame,

Because of your treatment within the FACT team of the GGZ Oost Brabant, you will shortly be asked to complete a number of questionnaires. The questionnaires are administered to everyone. The answers are used to map out your problem as well as possible and to give you the best possible treatment.

# Research:

Not so long ago, one of these questionnaires, the substance use questionnaire, was replaced. The questionnaire about substance use that is currently being used, the TAPS, has been used in America for some time, but is still new for the Netherlands. That is why we want to investigate how good this Dutch version is. We ask for your cooperation for this investigation. Your cooperation is voluntary, but we do need your written consent.

#### Participation:

If you participate, you can always change your mind and indicate that you no longer want to participate. You don't have to say why you're stopping. We will then not use your data in the research.

### What happens to your data?

In addition to the results of the TAPS and the supplementary questionnaire, we also want to include some other data in the study for this study. These are your gender, age, diagnosis and the results of other questionnaires you complete in connection with your FACT treatment. This allows us to better understand the role substance use plays, which helps us improve treatment.

To protect your privacy, your data are assigned with a code. Your name, and other information that may identify you as a person, will be omitted and replaced by this code. The data can only be traced back to you with the key of the code. This key is safely stored within the GGZ Oost Brabant. The data that is used only contains the code, and therefore not your name or other data that can be traced back to you. Also in reports and publications about this research, the data cannot be traced back to you.

We want to store your answers to all questionnaires in a computer file in the secure environment of the GGZ. The answers and your other data are entered by the researchers, who also have access to your file. The results of the extra questionnaire that is administered for this study must be kept for 15 years.

#### Informed consent form:

If you give permission, we will ask you to confirm this in writing on the corresponding declaration of consent. By your written consent, you indicate that you have understood the information and agree to participate in the study. Both you and the researcher will receive a signed version of this consent form.

Would you like to know more? Then you can call Birgit Seelen (telephone: 0492-844300).

Kind regards,

Birgit Seelen, GZ psychologist



### CONSENT FORM: Research into the TAPS questionnaire

- I've read the information letter. I could also ask questions. My questions have been sufficiently answered. I had plenty of time to decide whether to participate.
- I know that taking part is voluntary. I also know that I can decide at any time not to participate or to stop the study. I don't have to give a reason for that.
- I give permission for the collection and use of my answers to answer the research question in this study.
- I know that the researchers need my answers and some other data for this. I give the researchers permission to use this data.

Name of subject:

Signature: Date :\_\_/\_\_/\_\_

I declare that I have fully informed this subject about the said study.

Name investigator (or representative):

Signature: Date: \_\_/\_\_/\_\_

\* Strike out what does not apply.

I want to participate tot his research:

The subject receives a complete information letter, together with a signed version of the consent form